CLINICAL TRIAL: NCT02308748
Title: Five Period Crossover Study of the Ability of Late Sodium or Calcium Current Block (Mexiletine, Lidocaine, or Diltiazem) to Balance the Electrocardiographic Effects of hERG Potassium Current Block (Dofetilide or Moxifloxacin)
Brief Title: Ability of Late Sodium or Calcium Current Block to Balance the ECG Effects of Potassium Current Block
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Food and Drug Administration (FDA) (U.S. Federal Agency)
Collaborators: Spaulding Clinical Research LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 14-022D; SCR-003 (Other: Spaulding Clinical Research)
Record Dates: First submitted 2014-11-06; First posted 2014-12-04 (Estimated); Results first posted 2016-06-08 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Drug-induced QT Prolongation; Pharmacokinetics; Pharmacodynamics
MeSH Terms: interventions — dofetilide; Mexiletine; Lidocaine; Moxifloxacin; Diltiazem; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Dofetilide (Active Comparator): Dofetilide alone arm
  Interventions: Drug: Dofetilide
- Dofetilide + Mexiletine (Active Comparator): Dofetilide combined with mexiletine
  Interventions: Drug: Dofetilide; Drug: Mexiletine
- Dofetilide + Lidocaine (Active Comparator): Dofetilide combined with lidocaine
  Interventions: Drug: Dofetilide; Drug: Lidocaine
- Moxifloxacin + Diltiazem (Active Comparator): Moxifloxacin with and without diltiazem.
  Interventions: Drug: Moxifloxacin; Drug: Diltiazem
- Placebo (Placebo Comparator): Placebo (#2 gelcap and intravenous saline)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dofetilide — * 8 am: Placebo
  * 12 pm (noon): 250 µg
  * 5:30 pm: 250 µg
  Other Names: Tikosyn
  Arms: Dofetilide; Dofetilide + Lidocaine; Dofetilide + Mexiletine
Drug: Mexiletine — * 8 am: weight x 4 mg/kg
  * 12 pm (noon): Same as at 8 am
  * 5:30 pm: Same as at 8 am
  Other Names: Mexitil
  Arms: Dofetilide + Mexiletine
Drug: Lidocaine — * 9 am : 30 µg/min per kg (loading) for 60 minutes and 10 µg/min per kg (maintenance) for 30 minutes
  * 2 pm: 55 µg/min per kg (loading) for 60 minutes and 20 µg/min per kg (maintenance) for 30 minutes
  * 7:30 pm: 52 µg/min per kg (loading) for 60 minutes and 20 µg/min per kg (maintenance) for 30 minutes
  Other Names: Lidocaine hydrochloride
  Arms: Dofetilide + Lidocaine
Drug: Moxifloxacin — * 9 am: 5.63 mg/h per kg (loading) for 1 hour and 0.26 mg/h per kg (maintenance for 30 minutes)
  * 2 pm: 6.14 mg/h per kg (loading) for 1 hour and 0.49 mg/h per kg (maintenance for 30 minutes)
  * 7:30 pm: 2.23 mg/h per kg (loading) for 1 hour and 0.49 mg/h per kg (maintenance for 30 minutes)
  Other Names: Avelox
  Arms: Moxifloxacin + Diltiazem
Drug: Diltiazem — • 7:30 pm: 330 µg/h per kg (loading) for 60 minutes and 61 µg/h per kg (maintenance) for 30 minutes
  Other Names: Diltiazem hydrochloride
  Arms: Moxifloxacin + Diltiazem
Drug: Placebo — Placebo (#2 Gelcap or IV saline)
  Other Names: #2 Gelcaps or IV saline
  Arms: Placebo

SUMMARY:
The primary objective of this research study is to test the hypothesis that late sodium current blocking drugs (mexiletine or lidocaine) can attenuate the effect of hERG potassium channel blocking drugs (dofetilide) on ventricular repolarization (QTc) by shortening early repolarization (J-Tpeakc). The secondary object is to assess the ability of calcium channel block (diltiazem) to reduce the QTc prolongation associated with hERG block (moxifloxacin).

DETAILED DESCRIPTION:
This is a randomized, double-blind, 5-period crossover study in healthy male and female subjects, 18 to 35 years of age, to compare the electrophysiological response of hERG potassium channel blocking drugs with and without the addition of late sodium or calcium channel blocking drugs. The 5 treatment periods are 1) dofetilide alone, 2) mexiletine with and without dofetilide, 3) lidocaine with and without dofetilide, 4) moxifloxacin with and without diltiazem and 5) placebo. During each treatment period, 12 blood samples for pharmacokinetic measurements are obtained with matched 12-lead ECG recordings.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a healthy man or woman, 18 to 35 years of age, inclusive, who weighs at least 50 kg (110 pounds), no more than 85 kg (197 pounds) and has a body mass index of 18 to 27 kg/m2, inclusive, at Screening.
2. Subject has normal medical history findings, clinical laboratory results, vital sign measurements, 12 lead ECG results, and physical examination findings at Screening or, if abnormal, the abnormality is not considered clinically significant (as determined and documented by the investigator or designee).
3. Male or female subjects must agree to practice 2 highly effective methods of birth control (as determined by the investigator or designee; one of the methods must be a barrier technique) from Screening until 30 days after the last dose of study drug.

Exclusion Criteria:

* 1. Subject has a 12 lead safety ECG result at Screening or Check in of Period 1 with evidence of any of the following abnormalities:

  * QT corrected interval (QTc) using Fridericia correction (QTcF) >430 milliseconds (ms)
  * PR interval >220 ms or <120 ms
  * QRS duration >110 ms
  * Second- or third-degree atrioventricular block
  * Complete left or right bundle branch block or incomplete right bundle branch block
  * Heart rate <50 or >90 beats per minute
  * Pathological Q-waves (defined as Q wave >40 ms)
  * Ventricular pre-excitation

    2. Subject has more than 12 ectopic beats during the 3 hour Holter ECG at Screening.

    3. Subject has a history of unexplained syncope, structural heart disease, long QT syndrome, heart failure, myocardial infarction, angina, unexplained cardiac arrhythmia, torsades de pointes, ventricular tachycardia, or placement of a pacemaker or implantable defibrillator. Subjects will also be excluded if there is a family history of long QT syndrome (genetically proven or suggested by sudden death of a close relative due to cardiac causes at a young age) or Brugada syndrome.

    4. Subject has a history or current evidence of any clinically significant (as determined by the investigator) cardiovascular, dermatologic, endocrine, gastrointestinal, hematologic, hepatic, immunologic, metabolic, neurologic, psychiatric, pulmonary, renal, urologic, and/or other major disease or malignancy (excluding nonmelanoma skin cancer). The investigator may allow exceptions to these criteria (e.g., stable mild joint disease [that will not interfere with or influence the activities required by the protocol, in the opinion of the investigator], cholecystectomy, childhood asthma) following discussion with the medical monitor.

    5. Subject has a history of thoracic surgery.

    6. Subject has any condition possibly affecting study drug absorption (e.g., gastrectomy, Crohn's disease, irritable bowel syndrome).

    7. Subject has a skin condition likely to compromise ECG electrode placement.

    8. Subject is a female with breast implants.

    9. Subject's laboratory test results at Screening or Check in of Period 1 are outside the reference ranges provided by the clinical laboratory and considered clinically significant (as determined and documented by the investigator or designee).

    10. Subject's laboratory test results at Screening or Check in of Period 1 indicate hypokalemia, hypocalcemia, or hypomagnesemia according to lower limits of the reference ranges provided by the clinical laboratory.

    11. Subject's laboratory test results at Screening or Check in of Period 1 are >2 × the upper limit of normal (ULN) for alanine aminotransferase or aspartate aminotransferase, >1.5 × ULN for bilirubin, or >1.5 × ULN for creatinine.

    12. Subject has a positive test result at Screening for human immunodeficiency virus, hepatitis C antibodies, or hepatitis B surface antigen.

    13. Subject has a mean systolic blood pressure <90 or >140 mmHg or a mean diastolic blood pressure <50 or >90 mmHg at either Screening or Check in of Period 1.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2014-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Sanabria, MD, Principal Investigator — Spaulding Clinical

REFERENCES:
- [Result] Johannesen L, Vicente J, Mason JW, Erato C, Sanabria C, Waite-Labott K, Hong M, Lin J, Guo P, Mutlib A, Wang J, Crumb WJ, Blinova K, Chan D, Stohlman J, Florian J, Ugander M, Stockbridge N, Strauss DG. Late sodium current block for drug-induced long QT syndrome: Results from a prospective clinical trial. Clin Pharmacol Ther. 2016 Feb;99(2):214-23. doi: 10.1002/cpt.205. Epub 2015 Nov 28. PMID 26259627
- [Derived] Vicente J, Johannesen L, Hosseini M, Mason JW, Sager PT, Pueyo E, Strauss DG. Electrocardiographic Biomarkers for Detection of Drug-Induced Late Sodium Current Block. PLoS One. 2016 Dec 30;11(12):e0163619. doi: 10.1371/journal.pone.0163619. eCollection 2016. PMID 28036334
- [Derived] Johannesen L, Vicente J, Hosseini M, Strauss DG. Automated Algorithm for J-Tpeak and Tpeak-Tend Assessment of Drug-Induced Proarrhythmia Risk. PLoS One. 2016 Dec 30;11(12):e0166925. doi: 10.1371/journal.pone.0166925. eCollection 2016. PMID 28036330

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 44 healthy volunteers were assessed for eligibility. 15 subjects were excluded because they did not meet the inclusion criteria. 22 of 29 subjects who met the inclusion criteria were randomized and allocated to receive crossed-over intervention. Williams Latin square design balanced for first-order carryover effects was used for randomization.
Groups:
- A-D-E-C-B: All subjects received the same 5 treatments, separated by 6 days of washout, but were randomized to receive them in different orders. Subjects in this arm received them in the following order:
  Treatment A (dofetilide) Treatment D (moxifloxacin + diltiazem) Treatment E (placebo) Treatment C (dofetilide + mexiletine) Treatment B (dofetilide + lidocaine)
- B-C-E-D-A: All subjects received the same 5 treatments, separated by 6 days of washout, but were randomized to receive them in different orders. Subjects in this arm received them in the following order:
  Treatment B (dofetilide + lidocaine) Treatment C (dofetilide + mexiletine) Treatment E (placebo) Treatment D (moxifloxacin + diltiazem) Treatment A (dofetilide)
- C-D-B-A-E: All subjects received the same 5 treatments, separated by 6 days of washout, but were randomized to receive them in different orders. Subjects in this arm received them in the following order:
  Treatment C (dofetilide + mexiletine) Treatment D (moxifloxacin + diltiazem) Treatment B (dofetilide + lidocaine) Treatment A (dofetilide) Treatment E (placebo)
- D-C-A-B-E: All subjects received the same 5 treatments, separated by 6 days of washout, but were randomized to receive them in different orders. Subjects in this arm received them in the following order:
  Treatment D (moxifloxacin + diltiazem) Treatment C (dofetilide + mexiletine) Treatment A (dofetilide) Treatment B (dofetilide + lidocaine) Treatment E (placebo)
- E-A-B-D-C: All subjects received the same 5 treatments, separated by 6 days of washout, but were randomized to receive them in different orders. Subjects in this arm received them in the following order:
  Treatment E (placebo) Treatment A (dofetilide) Treatment B (dofetilide + lidocaine) Treatment D (moxifloxacin + diltiazem) Treatment C (dofetilide + mexiletine)
- D-A-C-E-B: All subjects received the same 5 treatments, separated by 6 days of washout, but were randomized to receive them in different orders. Subjects in this arm received them in the following order:
  Treatment D (moxifloxacin + diltiazem) Treatment A (dofetilide) Treatment C (dofetilide + mexiletine) Treatment E (placebo) Treatment B (dofetilide + lidocaine)
- E-B-A-C-D: All subjects received the same 5 treatments, separated by 6 days of washout, but were randomized to receive them in different orders. Subjects in this arm received them in the following order:
  Treatment E (placebo) Treatment B (dofetilide + lidocaine) Treatment A (dofetilide) Treatment C (dofetilide + mexiletine) Treatment D (moxifloxacin + diltiazem)
- A-E-D-B-C: All subjects received the same 5 treatments, separated by 6 days of washout, but were randomized to receive them in different orders. Subjects in this arm received them in the following order:
  Treatment A (dofetilide) Treatment E (placebo) Treatment D (moxifloxacin + diltiazem) Treatment B (dofetilide + lidocaine) Treatment C (dofetilide + mexiletine)
- B-E-C-A-D: All subjects received the same 5 treatments, separated by 6 days of washout, but were randomized to receive them in different orders. Subjects in this arm received them in the following order:
  Treatment B (dofetilide + lidocaine) Treatment E (placebo) Treatment C (dofetilide + mexiletine) Treatment A (dofetilide) Treatment D (moxifloxacin + diltiazem)
- C-B-D-E-A: All subjects received the same 5 treatments, separated by 6 days of washout, but were randomized to receive them in different orders. Subjects in this arm received them in the following order:
  Treatment C (dofetilide + mexiletine) Treatment B (dofetilide + lidocaine) Treatment D (moxifloxacin + diltiazem) Treatment E (placebo) Treatment A (dofetilide)
Period: Period 1
Arm/Group | A-D-E-C-B | B-C-E-D-A | C-D-B-A-E | D-C-A-B-E | E-A-B-D-C | D-A-C-E-B | E-B-A-C-D | A-E-D-B-C | B-E-C-A-D | C-B-D-E-A
Started | 2 | 2 | 2 | 2 | 2 | 3 | 2 | 2 | 2 | 3
Completed | 2 | 2 | 1 (One subject withdraw consent before starting Period 2) | 2 | 2 | 3 | 2 | 2 | 2 | 3
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | A-D-E-C-B | B-C-E-D-A | C-D-B-A-E | D-C-A-B-E | E-A-B-D-C | D-A-C-E-B | E-B-A-C-D | A-E-D-B-C | B-E-C-A-D | C-B-D-E-A
Started | 2 | 2 | 1 | 2 | 2 | 3 | 2 | 2 | 2 | 3
Completed | 2 | 2 | 1 | 2 | 2 | 3 | 2 | 1 | 2 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Period: Period 3
Arm/Group | A-D-E-C-B | B-C-E-D-A | C-D-B-A-E | D-C-A-B-E | E-A-B-D-C | D-A-C-E-B | E-B-A-C-D | A-E-D-B-C | B-E-C-A-D | C-B-D-E-A
Started | 2 | 2 | 1 | 2 | 2 | 3 | 2 | 1 | 2 | 3
Completed | 2 | 2 | 1 | 2 | 2 | 3 | 2 | 1 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Period 4
Arm/Group | A-D-E-C-B | B-C-E-D-A | C-D-B-A-E | D-C-A-B-E | E-A-B-D-C | D-A-C-E-B | E-B-A-C-D | A-E-D-B-C | B-E-C-A-D | C-B-D-E-A
Started | 2 | 2 | 1 | 2 | 2 | 3 | 2 | 1 | 2 | 2
Completed | 2 | 2 | 1 | 2 | 2 | 3 | 2 | 1 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 5
Arm/Group | A-D-E-C-B | B-C-E-D-A | C-D-B-A-E | D-C-A-B-E | E-A-B-D-C | D-A-C-E-B | E-B-A-C-D | A-E-D-B-C | B-E-C-A-D | C-B-D-E-A
Started | 2 | 2 | 1 | 2 | 2 | 3 | 2 | 1 | 2 | 2
Completed | 1 | 2 | 1 | 2 | 2 | 3 | 2 | 1 | 1 | 2
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants who were randomized to receive either dofetilide alone, dofetilide + mexiletine, dofetilide + lidocaine, moxifloxacin + diltiazem or placebo.
Arm/Group | All Study Participants
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.1 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 22
Weight [Mean (Standard Deviation); unit: kg] | 69.9 (9.0)
Systolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 109.5 (5.5)
Diastolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 60.2 (3.5)
Heart rate [Mean (Standard Deviation); unit: beats per minute (bpm)] | 61.3 (6.7)
PR interval [Mean (Standard Deviation); unit: ms] | 160.8 (19.1)
QRS duration [Mean (Standard Deviation); unit: ms] | 86.7 (8.5)
J-Tpeakc (heart rate corrected J-Tpeak interval) [Mean (Standard Deviation); unit: ms] | 229.5 (19.0)
Tpeak-Tend interval [Mean (Standard Deviation); unit: ms] | 81.9 (6.4)
QTc (Fridericia's heart rate corrected QT interval) [Mean (Standard Deviation); unit: ms] | 397.8 (14.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Placebo Corrected Change From Baseline QTc and J-Tpeakc Intervals on the ECG Measured in Milliseconds When Dofetilide is Administered With Mexiletine or Lidocaine Compared to When Dofetilide is Administered Alone at Evening Dose on Treatment Day
Description: After 3rd dose of mexiletine or lidocaine (evening dose) on treatment day when combined with dofetilide to evening dose on dofetilide alone day.
Time Frame: 5 weeks
Population: All study participants that completed placebo and dofetilide alone as well as dofetilide + mexiletine and/or dofetilide + lidocaine
Measure: Mean (95% Confidence Interval); unit: ms
Groups:
- Dofetilide Alone: Subjects that completed placebo and dofetilide alone interventions
- Dofetilide + Mexiletine: Subjects that completed placebo and dofetilide + mexiletine interventions
- Dofetilide + Lidocaine: Subjects that completed placebo and dofetilide + lidocaine interventions
Arm/Group | Dofetilide Alone | Dofetilide + Mexiletine | Dofetilide + Lidocaine
Number analyzed (Participants) | 20 | 20 | 18
ms
  Placebo corrected change from baseline in QTc | 37.9 [32.6 to 43.1] | 20.4 [15.1 to 25.6] | 18 [12.7 to 23.3]
  Placebo corrected change from baseline in J-Tpeakc | 24.0 [19.2 to 28.9] | 0.8 [-4.0 to 5.6] | 3.5 [-1.4 to 8.4]
Statistical Analysis 1: Comparison: Dofetilide Alone vs Dofetilide + Mexiletine; Change in QTc interval on the ECG measured in milliseconds when dofetilide is administered with mexiletine compared to when dofetilide is administered alone at evening dose on treatment day; Test type: Superiority or Other; p = 0.025, Mixed Models Analysis — Adjustment for multiple comparisons was performed according to the Bonferroni method; Mean Difference (Final Values) = -19.8, 95% CI 2-sided [-25.2 to -14.3]
Statistical Analysis 2: Comparison: Dofetilide Alone vs Dofetilide + Lidocaine; Change in QTc interval on the ECG measured in milliseconds when dofetilide is administered with lidocaine compared to when dofetilide is administered alone at evening dose on treatment day; Test type: Superiority or Other; p = 0.025, Mixed Models Analysis — Adjustment for multiple comparisons was performed according to the Bonferroni method; Mean Difference (Final Values) = -19.7, 95% CI 2-sided [-25.2 to -14.1]
Statistical Analysis 3: Comparison: Dofetilide Alone vs Dofetilide + Mexiletine; Change in J-Tpeakc interval on the ECG measured in milliseconds when dofetilide is administered with mexiletine compared to when dofetilide is administered alone at evening dose on treatment day; Test type: Superiority or Other; p = 0.025, Mixed Models Analysis — Adjustment for multiple comparisons was performed according to the Bonferroni method; Mean Difference (Final Values) = -23.2, 95% CI 2-sided [-28.0 to -18.3]
Statistical Analysis 4: Comparison: Dofetilide Alone vs Dofetilide + Lidocaine; Change in J-Tpeakc interval on the ECG measured in milliseconds when dofetilide is administered with lidocaine compared to when dofetilide is administered alone at evening dose on treatment day; Test type: Superiority or Other; p = 0.025, Mixed Models Analysis — Adjustment for multiple comparisons was performed according to the Bonferroni method; Mean Difference (Final Values) = -20.5, 95% CI 2-sided [-25.5 to -15.5]

2. Secondary Outcome: Change in Placebo Corrected Change From Baseline QTc Interval on the ECG Measured in Milliseconds When Moxifloxacin is Administered With Diltiazem at the Evening Dose Compared to When Moxifloxacin is Administered Alone at Afternoon Dose on Treatment Day.
Description: Evening dose (moxifloxacin+diltiazem) versus afternoon dose (diltiazem alone).
Time Frame: 5 weeks
Population: All study participants that completed placebo, moxifloxacin and moxifloxacin + diltiazem
Measure: Mean (95% Confidence Interval); unit: ms
Groups:
- Moxifloxacin Alone: Subjects that completed placebo and moxifloxacin alone interventions
- Moxifloxacin + Diltiazem: Subjects that completed placebo and moxifloxacin + diltiazem interventions
Arm/Group | Moxifloxacin Alone | Moxifloxacin + Diltiazem
Number analyzed (Participants) | 19 | 19
ms | 29.9 [24.6 to 35.2] | 31.3 [26.0 to 36.6]
Statistical Analysis 1: Comparison: Moxifloxacin Alone vs Moxifloxacin + Diltiazem; Test type: Superiority or Other; p = 0.025, Mixed Models Analysis — Adjustment for multiple comparisons was performed according to the Bonferroni method; Mean Difference (Final Values) = 2.9, 95% CI 2-sided [-1 to 6.7]

ADVERSE EVENTS:
Groups:
- Dofetilide: Dofetilide alone arm
  Dofetilide: • 8 am: Placebo
  * 12 pm (noon): 250 µg
  * 5:30 pm: 250 µg
- Dofetilide + Lidocaine: Dofetilide combined with lidocaine
  Dofetilide: • 8 am: Placebo
  * 12 pm (noon): 250 µg
  * 5:30 pm: 250 µg
  Lidocaine: • 9 am : 30 µg/min per kg (loading) for 60 minutes and 10 µg/min per kg (maintenance) for 30 minutes
  * 2 pm: 55 µg/min per kg (loading) for 60 minutes and 20 µg/min per kg (maintenance) for 30 minutes
  * 7:30 pm: 52 µg/min per kg (loading) for 60 minutes and 20 µg/min per kg (maintenance) for 30 minutes
- Dofetilide + Mexiletine: Dofetilide combined with mexiletine
  Dofetilide: • 8 am: Placebo
  * 12 pm (noon): 250 µg
  * 5:30 pm: 250 µg
  Mexiletine: • 8 am: weight x 4 mg/kg
  * 12 pm (noon): Same as at 8 am
  * 5:30 pm: Same as at 8 am
- Moxifloxacin + Diltiazem: Moxifloxacin with and without diltiazem.
  Moxifloxacin: • 9 am: 5.63 mg/h per kg (loading) for 1 hour and 0.26 mg/h per kg (maintenance for 30 minutes)
  * 2 pm: 6.14 mg/h per kg (loading) for 1 hour and 0.49 mg/h per kg (maintenance for 30 minutes)
  * 7:30 pm: 2.23 mg/h per kg (loading) for 1 hour and 0.49 mg/h per kg (maintenance for 30 minutes)
  Diltiazem: • 7:30 pm: 330 µg/h per kg (loading) for 60 minutes and 61 µg/h per kg (maintenance) for 30 minutes
Arm/Group | Dofetilide | Dofetilide + Lidocaine | Dofetilide + Mexiletine | Moxifloxacin + Diltiazem | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19 | 0/21 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 3/20 | 1/19 | 11/21 | 6/20 | 3/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dofetilide (N=20) | Dofetilide + Lidocaine (N=19) | Dofetilide + Mexiletine (N=21) | Moxifloxacin + Diltiazem (N=20) | Placebo (N=20)
Dizzines (Nervous system disorders) | 1 (1) | 1 (1) | 6 (6) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 | 4 (4) | 3 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 | 1 (1) | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No